CLINICAL TRIAL: NCT02577848
Title: Effects of Liraglutide on Left Ventricular Function in Patients With Non-ST-Segment Elevation Myocardial Infarction
Brief Title: GLP-1 on Non-ST-Segment Elevation Myocardial Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Chen Wei Ren, MD, Investigator, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLP-1-301xnk
Record Dates: First submitted 2015-10-15; First posted 2015-10-16 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Myocardial Infarction
Keywords: Glucagon-like peptide-1; Non-ST-segment elevation myocardial infarction; Left ventricular ejection fraction
MeSH Terms: conditions — Myocardial Infarction | interventions — Glucagon-Like Peptide 1; Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GLP-1 group (Experimental): liraglutide (Novo Nordisk, Bagsværd, Denmark); the frequency: Subcutaneous liraglutide were taken daily; duration: 7 days. After admission, the patients were treated with 0.6 mg liraglutide once daily for 2 day, then 1.2 mg liraglutide for another 2 day, and then 1.8 mg liraglutide for 3 days.
  Interventions: Drug: GLP-1
- placebo (Placebo Comparator): placebo (Novo Nordisk, Bagsværd, Denmark); the frequency: Placebo were taken daily; duration: After admission, the patients were treated with 0.6 mg placebo once daily for 2 day, then 1.2 mg placebo for another 2 day, and then 1.8 mg placebo for 3 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLP-1 — GLP-1 were taken daily for 7 days
  Other Names: Liraglutide
  Arms: GLP-1 group
Drug: Placebo — Placebo were taken daily for 7 days
  Arms: placebo

SUMMARY:
The investigators planned to evaluate the effects of liraglutide on left ventricular function in patients with non-ST-segment elevation myocardial infarction (NSTEMI).

DETAILED DESCRIPTION:
Patients with non-ST-segment elevation myocardial infarction (NSTEMI) are a heterogeneous group with respect to the risk of having a major adverse cardiac event (MACE). Elevation of blood glucose is a common metabolic disorder among patients with acute myocardial infarction (AMI) and is associated with adverse prognosis. Glucagon-like peptide-1 (GLP-1) is an incretin hormone that regulates plasma glucose. GLP-1 analogues have significant cardiovascular protective effects in patients with AMI. GLP-1 may have antioxidant and anti-inflammatory properties, and protect endothelial function. Studies in conscious, chronically instrumented dogs demonstrated that GLP-1 infusion increases insulin sensitivity and myocardial glucose uptake in postischemic contractile dysfunction and dilated cardiomyopathy. Liraglutide, a GLP-1 analogue, was reported to reduce cardiac rupture and infarct size and improve cardiac output in normal and diabetic mice. Continuous infusion of GLP-1 (1.5 pmol/kg/min) has been shown to improve functional recovery in patients with AMI complicated by decreased left ventricular function GLP-1 could protect against ischemia-reperfusion injury and improve cardiac function in patients with acute ST-segment elevation myocardial infarction. However, the effects of GLP-1 on NSTEMI patients remain unclear. The aim of this study was to evaluate the effects of liraglutide on left ventricular function in patients with NSTEMI.

ELIGIBILITY:
Inclusion Criteria:

non-ST-segment elevation myocardial infarction (NSTEMI )

Exclusion Criteria:

1. unconscious at presentation
2. had ST-segment elevation acute myocardial infarction
3. NSTEMI requiring emergency percutaneous coronary angiography
4. valvular heart disease
5. cardiogenic shock
6. hypoglycaemia
7. diabetic ketoacidosis
8. had a history of myocardial infarction
9. stent implantation
10. renal insufficiency
11. had previously undergone coronary artery bypass surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
left ventricular ejection fractions | at 3 months
  The primary efficacy endpoint was the effect of liraglutide on left ventricular ejection fractions (LVEF) measured by transthoracic echocardiography at 3 months .

SECONDARY OUTCOMES:
6-minute walk distance | at 3 months
  The change in6-minute walk distance at 3 months after treatment.
treatment-emergent adverse events | at 3 months
  Treatment-emergent adverse events (TEAEs): hypoglycaemia, pancreatitis, thyroid cancer

CONTACTS AND LOCATIONS:
Overall Officials: zhu Chen, Principal Investigator — World Health Organization
Locations (1):
- PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Montalescot G, Bolognese L, Dudek D, Goldstein P, Hamm C, Tanguay JF, ten Berg JM, Miller DL, Costigan TM, Goedicke J, Silvain J, Angioli P, Legutko J, Niethammer M, Motovska Z, Jakubowski JA, Cayla G, Visconti LO, Vicaut E, Widimsky P; ACCOAST Investigators. Pretreatment with prasugrel in non-ST-segment elevation acute coronary syndromes. N Engl J Med. 2013 Sep 12;369(11):999-1010. doi: 10.1056/NEJMoa1308075. Epub 2013 Sep 1. PMID 23991622
- [Background] Aronson D, Hammerman H, Kapeliovich MR, Suleiman A, Agmon Y, Beyar R, Markiewicz W, Suleiman M. Fasting glucose in acute myocardial infarction: incremental value for long-term mortality and relationship with left ventricular systolic function. Diabetes Care. 2007 Apr;30(4):960-6. doi: 10.2337/dc06-1735. PMID 17392556
- [Background] Lonborg J, Vejlstrup N, Kelbaek H, Botker HE, Kim WY, Mathiasen AB, Jorgensen E, Helqvist S, Saunamaki K, Clemmensen P, Holmvang L, Thuesen L, Krusell LR, Jensen JS, Kober L, Treiman M, Holst JJ, Engstrom T. Exenatide reduces reperfusion injury in patients with ST-segment elevation myocardial infarction. Eur Heart J. 2012 Jun;33(12):1491-9. doi: 10.1093/eurheartj/ehr309. Epub 2011 Sep 14. PMID 21920963
- [Background] Ceriello A, Novials A, Ortega E, Canivell S, La Sala L, Pujadas G, Esposito K, Giugliano D, Genovese S. Glucagon-like peptide 1 reduces endothelial dysfunction, inflammation, and oxidative stress induced by both hyperglycemia and hypoglycemia in type 1 diabetes. Diabetes Care. 2013 Aug;36(8):2346-50. doi: 10.2337/dc12-2469. Epub 2013 Apr 5. PMID 23564922
- [Background] Nikolaidis LA, Doverspike A, Hentosz T, Zourelias L, Shen YT, Elahi D, Shannon RP. Glucagon-like peptide-1 limits myocardial stunning following brief coronary occlusion and reperfusion in conscious canines. J Pharmacol Exp Ther. 2005 Jan;312(1):303-8. doi: 10.1124/jpet.104.073890. Epub 2004 Sep 8. PMID 15356213